CLINICAL TRIAL: NCT01894178
Title: STUDY EVALUATING THE PARKER-FLEX ENDOTRACHEAL TUBE FOR FIBEROPTIC INTUBATION ON OBESE PATIENTS
Brief Title: Study Examining Parker-Flex Endotracheal Tube for Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Lee Chang, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-31550
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parker Flex-Tip® Tracheal Tube (Active Comparator): Intubation of obese patients with the Parker Flex-Tip® Tracheal Tube
  Interventions: Device: Parker Flex-Tip® tracheal tube
- Portex® Tracheal Tube (Active Comparator): Intubation of obese patients with the Portex® Tracheal Tube
  Interventions: Device: Portex® Tracheal Tube

INTERVENTIONS:
Device: Parker Flex-Tip® tracheal tube
  Arms: Parker Flex-Tip® Tracheal Tube
Device: Portex® Tracheal Tube
  Arms: Portex® Tracheal Tube

SUMMARY:
A recent article examined the use of Parker Flex-Tip tubes to standard ETTs for oral fiberoptic intubation and concluded that there was a significant benefit in terms of difficulty encountered when using the Parker Flex-Tip. The Parker Flex-Tip tracheal tube has a flexible, curved, and tapered tip design different from traditional endotracheal tubes. The design allows the tube to lie closely against the fiberoptic scope that is often used to facilitate intubation, resulting in a smaller gap between the ETT and the fiberoptic scope. This may allow the ETT to clear anatomic obstructions more easily. The patients they examined had an average body mass index (BMI) categorized as normal weight. To our knowledge, there have not been any studies that have investigated the use of the Parker Flex-Tube for fiberoptic intubations in patients categorized as obese by BMI. Our hypothesis is that the Parker Flex-Tip ETT results in easier passage of the ETT over a fiberoptic scope during elective fiberoptic intubation of obese patients in comparison to a traditional ETT.

DETAILED DESCRIPTION:
This is a randomized, double-blinded study. Neither the patient nor the anesthesia practitioner advancing the ETT will know the group to which the patient has been assigned. On the day of surgery, participants will be randomized 1:1 to one of two groups. Both groups will be electively intubated with a fiberoptic scope. One group will be intubated using a Parker-Flex endotracheal tube and the second group of will be intubated with a standard endotracheal tube. There will be an equal probability of being assigned to either group. No placebo or control group will be used. Randomization will be computer-generated and assignments will be enclosed in sealed envelopes to provide allocation concealment. The anesthesiology technician involved in the case will open the envelope at the start of the case and will not be blinded to the study, due to the fact that the technician must prepare the endotracheal tube for the fiberoptic intubation.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 30 or greater
* American Society of Anesthesiologists (ASA) Physical Status Classification I- III
* Patients scheduled for elective procedures requiring general anesthesia and endotracheal intubation.

Exclusion Criteria:

* Predicted difficult airway based on physical exam and patient's history
* Rapid sequence intubation indicated (patients who require to be intubated as quickly as possible)
* Prior trauma or surgery in the oropharynx/larynx
* Known abnormal laryngeal structures (tumors)
* Infectious and toxic conditions
* Cervical spine instability
* Emergency surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Parker Flex-Tip® Tracheal Tube: Intubation of obese patients with the Parker Flex-Tip® Tracheal Tube
  Parker Flex-Tip® tracheal tube
- Portex® Tracheal Tube: Intubation of obese patients with the Portex® Tracheal Tube
  Portex® Tracheal Tube
Period: Overall Study
Arm/Group | Parker Flex-Tip® Tracheal Tube | Portex® Tracheal Tube
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parker Flex-Tip® Tracheal Tube | Portex® Tracheal Tube | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Length of Time Required for Successful Advancement of Endotracheal Tube Into Trachea
Time Frame: following successful intubation or lasting longer than 120 seconds
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Parker Flex-Tip® Tracheal Tube | Portex® Tracheal Tube
Number analyzed (Participants) | 30 | 30
seconds | 6.36 [5 to 10.4] | 8.81 [5.3 to 14.2]

2. Secondary Outcome: Percentage of Endotracheal Intubations Successful on First Attempt Attempts
Time Frame: following successful intubation or more than 5 attempts
Measure: Number; unit: percentage of successful first attempts
Arm/Group | Parker Flex-Tip® Tracheal Tube | Portex® Tracheal Tube
Number analyzed (Participants) | 30 | 30
percentage of successful first attempts | 62 | 73

3. Other Pre Specified Outcome: Number of Failed Attempts of Placing Endotracheal Tube Into Trachea
Description: The intent is to report the number of attempts required to successfully advance the endotracheal tube into the trachea.
Time Frame: following intubation attempt
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Parker Flex-Tip® Tracheal Tube | Portex® Tracheal Tube
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No